CLINICAL TRIAL: NCT04392960
Title: Molecular, Magnetic Resonance, and Echocardiographic Imaging Combined With Biomarkers of Cardiac and Clonal Disease to Predict Survival and Assess Response to Therapy in Cardiac AL Amyloidosis
Brief Title: Novel Imaging Tools in Newly-diagnosed Patients With Cardiac AL Amyloidosis
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Fondazione IRCCS Policlinico San Matteo di Pavia (Other)
Responsible Party: Principal Investigator, Giovanni Palladini, Principal Investigator, Fondazione IRCCS Policlinico San Matteo di Pavia
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: AC-015-IT
Record Dates: First submitted 2020-02-27; First posted 2020-05-19 (Actual); Last update posted 2025-05-07 (Actual); Status verified 2025-05

CONDITIONS: AL Amyloidosis
Keywords: Amyloidosis; Prognosis; [18F]Florbetaben
MeSH Terms: conditions — Immunoglobulin Light-chain Amyloidosis; Amyloidosis | interventions — 4-(N-methylamino)-4'-(2-(2-(2-fluoroethoxy)ethoxy)ethoxy)stilbene

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- 18F-florbetaben PET-CT scans (Experimental)
  Interventions: Drug: [18F]Florbetaben

INTERVENTIONS:
Drug: [18F]Florbetaben — Patients will undergo on the same day:
  * 18F-florbetaben PET-CT scans. The dose to be injected intravenously (6 second/mL) will be 370 MBq (for a 70 Kg patient);
  * standard assessment of clonal and organ disease;
  * echocardiography;
  * cardiac magnetic resonance.
  All the patients will undergo those evaluations at baseline and 6 months after treatment initiation.

SUMMARY:
This will be a systematic, combined, prospective assessment of the novel echographic, CMR, and PET imaging tools in newly-diagnosed patients with cardiac AL amyloidosis at baseline and after treatment.

ELIGIBILITY:
Inclusion Criteria:

* age more than 18;
* histological diagnosis of AL amyloidosis;
* measurable cardiac involvement as per current response criteria (i.e. NT-proBNP >650 ng/L);
* measurable hematologic disease (dFLC >20 mg/L);
* adequate renal function (eGFR >30 mL/min) in order to be safely administered gadolinium;
* absence of atrial fibrillation with uncontrolled heart rate;
* absence of implantable cardiac devices;
* absence of pulmonary amyloidosis histologically documented;
* plan to start anti-plasma cell chemotherapy;
* plan to assess response at the Pavia center after 6 months;
* have given written informed consent to participate.

Exclusion Criteria:

* non-AL amyloidosis;
* NYHA class IV;
* PS-ECOG >3;
* severe allergy to paramagnetic tracer;
* severe claustrophobia;
* pregnant or nursing women;

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 69 (Estimated)
Dates: Start 2020-07-22 (Actual); Primary Completion 2025-06-30 (Estimated); Study Completion 2025-06-30 (Estimated)

PRIMARY OUTCOMES:
Evaluation of the prognostic relevance of advanced imaging variables. | 12 months after diagnosis
  - for CMR: T1, T2, ECV, indexed volumes, mass, ejection fraction (EF);
Evaluation of the prognostic relevance of advanced imaging variables. | 12 months after diagnosis
  - for echocardiography: left ventricular wall thickness (mLVW), EF, 2D-GLS, midwall fractional shortening (mFS), and stroke volume index (SVI);
Evaluation of the prognostic relevance of advanced imaging variables. | 12 months after diagnosis
  - for F-PET: myocardial uptake score.
Evaluation of advanced imaging variables in response assessment. | 6 months after initiation of chemotherapy targeting the amyloid plasma cell clone
  The same variables considered at baseline will be measured 6 months after initiation of chemotherapy targeting the amyloid plasma cell clone. Changes in these variables compared to baseline will be considered.

CONTACTS AND LOCATIONS:
Locations (1):
- Fondazione IRCCS Policlinico San Matteo, Pavia, Italy

REFERENCES:
- [Background] Palladini G, Barassi A, Klersy C, Pacciolla R, Milani P, Sarais G, Perlini S, Albertini R, Russo P, Foli A, Bragotti LZ, Obici L, Moratti R, Melzi d'Eril GV, Merlini G. The combination of high-sensitivity cardiac troponin T (hs-cTnT) at presentation and changes in N-terminal natriuretic peptide type B (NT-proBNP) after chemotherapy best predicts survival in AL amyloidosis. Blood. 2010 Nov 4;116(18):3426-30. doi: 10.1182/blood-2010-05-286567. Epub 2010 Jul 19. PMID 20644111
- [Background] Dispenzieri A, Gertz MA, Kyle RA, Lacy MQ, Burritt MF, Therneau TM, Greipp PR, Witzig TE, Lust JA, Rajkumar SV, Fonseca R, Zeldenrust SR, McGregor CG, Jaffe AS. Serum cardiac troponins and N-terminal pro-brain natriuretic peptide: a staging system for primary systemic amyloidosis. J Clin Oncol. 2004 Sep 15;22(18):3751-7. doi: 10.1200/JCO.2004.03.029. PMID 15365071
- [Background] Wechalekar AD, Schonland SO, Kastritis E, Gillmore JD, Dimopoulos MA, Lane T, Foli A, Foard D, Milani P, Rannigan L, Hegenbart U, Hawkins PN, Merlini G, Palladini G. A European collaborative study of treatment outcomes in 346 patients with cardiac stage III AL amyloidosis. Blood. 2013 Apr 25;121(17):3420-7. doi: 10.1182/blood-2012-12-473066. Epub 2013 Mar 11. PMID 23479568
- [Background] Palladini G, Lavatelli F, Russo P, Perlini S, Perfetti V, Bosoni T, Obici L, Bradwell AR, D'Eril GM, Fogari R, Moratti R, Merlini G. Circulating amyloidogenic free light chains and serum N-terminal natriuretic peptide type B decrease simultaneously in association with improvement of survival in AL. Blood. 2006 May 15;107(10):3854-8. doi: 10.1182/blood-2005-11-4385. Epub 2006 Jan 24. PMID 16434487
- [Background] Palladini G, Dispenzieri A, Gertz MA, Kumar S, Wechalekar A, Hawkins PN, Schonland S, Hegenbart U, Comenzo R, Kastritis E, Dimopoulos MA, Jaccard A, Klersy C, Merlini G. New criteria for response to treatment in immunoglobulin light chain amyloidosis based on free light chain measurement and cardiac biomarkers: impact on survival outcomes. J Clin Oncol. 2012 Dec 20;30(36):4541-9. doi: 10.1200/JCO.2011.37.7614. Epub 2012 Oct 22. PMID 23091105
- [Background] Mishra S, Guan J, Plovie E, Seldin DC, Connors LH, Merlini G, Falk RH, MacRae CA, Liao R. Human amyloidogenic light chain proteins result in cardiac dysfunction, cell death, and early mortality in zebrafish. Am J Physiol Heart Circ Physiol. 2013 Jul 1;305(1):H95-103. doi: 10.1152/ajpheart.00186.2013. Epub 2013 Apr 26. PMID 23624626
- [Background] Diomede L, Rognoni P, Lavatelli F, Romeo M, del Favero E, Cantu L, Ghibaudi E, di Fonzo A, Corbelli A, Fiordaliso F, Palladini G, Valentini V, Perfetti V, Salmona M, Merlini G. A Caenorhabditis elegans-based assay recognizes immunoglobulin light chains causing heart amyloidosis. Blood. 2014 Jun 5;123(23):3543-52. doi: 10.1182/blood-2013-10-525634. Epub 2014 Mar 24. PMID 24665135
- [Background] Weiss BM, Wong SW, Comenzo RL. Beyond the plasma cell: emerging therapies for immunoglobulin light chain amyloidosis. Blood. 2016 May 12;127(19):2275-80. doi: 10.1182/blood-2015-11-681650. Epub 2016 Feb 23. PMID 26907632
- [Background] Barros-Gomes S, Williams B, Nhola LF, Grogan M, Maalouf JF, Dispenzieri A, Pellikka PA, Villarraga HR. Prognosis of Light Chain Amyloidosis With Preserved LVEF: Added Value of 2D Speckle-Tracking Echocardiography to the Current Prognostic Staging System. JACC Cardiovasc Imaging. 2017 Apr;10(4):398-407. doi: 10.1016/j.jcmg.2016.04.008. Epub 2016 Sep 14. PMID 27639764
- [Background] Fontana M, Banypersad SM, Treibel TA, Abdel-Gadir A, Maestrini V, Lane T, Gilbertson JA, Hutt DF, Lachmann HJ, Whelan CJ, Wechalekar AD, Herrey AS, Gillmore JD, Hawkins PN, Moon JC. Differential Myocyte Responses in Patients with Cardiac Transthyretin Amyloidosis and Light-Chain Amyloidosis: A Cardiac MR Imaging Study. Radiology. 2015 Nov;277(2):388-97. doi: 10.1148/radiol.2015141744. Epub 2015 May 21. PMID 25997029